CLINICAL TRIAL: NCT01267214
Title: The Efficacy and Safety of Intraarticular Sodium Hyaluronate (Hyalgan) After Proximal Tibial Osteotomy in Treatment of Knee Osteoarthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TRB Chemedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGN-THA-08-01
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid; Osteotomy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Osteotomy plus Hyalgan (Experimental): Osteotomy at Week 0 Hyalgan injection at Week 2, 3, 4, 5, 6, 24, 25, 26, 27, 28
  Interventions: Drug: Sodium Hyaluronate (Hyalgan)
- Osteotomy alone (Other)
  Interventions: Procedure: Osteotomy alone

INTERVENTIONS:
Drug: Sodium Hyaluronate (Hyalgan) — 1% Sodium Hyaluronate in prefilled syringe
  Arms: Osteotomy plus Hyalgan
Procedure: Osteotomy alone — no injection
  Arms: Osteotomy alone

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Hyalgan after proximal tibial osteotomy in treatment of knee osteoarthritis patients. Normally, OA patients who were treated with osteotomy will not be treated with any SYSADOA after operation, even though their cartilage's not completely loss, so osteotomy plus HA injection should provide more benefit to patients than osteotomy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 35 and 65 years with primary knee OA with malalignment
2. Mild to moderate OA of grade II or III severity on the Kellgren-Lawrence scale with require treatment by osteotomy
3. Malalignment is not exceed 15 degree (+,-)
4. Pain on walking (15 m) ≥ 40 mm.
5. Range of motion > 90 degree
6. Evidence of adequate contraceptive methods in women of childbearing age

Exclusion Criteria:

1. Previous surgery on affected knee
2. Previous intraarticular intervention within the last 3 months (eg. Steroid, anaesthetic, Sodium hyaluronate)
3. Oral SYSADOA treatment (chondroitin, glucosamine, diacerein) within 2 months prior to study start
4. Known or suspected infection of the affected joint
5. Painful knee condition due to another cause than chondral lesions, such as Sudeck's atrophy, intraarticular neoplasm, pigmented villonodular synovitis, chondromatosis
6. Poor general health or other conditions which would make regular hospital attendance difficult
7. Ascertained hypersensitivity to any component used in the study (eg. Hyaluronic acid, diclofenac, morphine, omeprazole and paracetamol)
8. Hypersensitivity to avian protein
9. Ongoing or previous participation in a clinical study within the last 3 months

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Joint Space Width | 12 months
Global assessment | 12 months
  assess by Patient and investigator
WOMAC section A, B, C | 12 months
  Pain score
Rescue medicine consumption | 12 months
  Diclofenac consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Faculty of Medicine, Mahidol university, Bangkok, Bangkok, Thailand